CLINICAL TRIAL: NCT02320682
Title: Bone Metabolism Adjacent to Hip Prosthetic Surfaces. A Randomized Clinical F-PET/CT Study.
Brief Title: Bone Metabolism Adjacent to Hip Prosthetic Surfaces. A Clinical F-PET/CT Study
Acronym: Fp-III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: gosta ullmark (Other)
Responsible Party: Sponsor-Investigator, gosta ullmark, Assistent Professor, Uppsala University
Organization: Uppsala University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fingerprint III
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Hip Osteo Arthritis
MeSH Terms: interventions — Surgical Procedures, Operative; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exeter femur component and Delta TT acetabular component (Active Comparator)
  Interventions: Device: Surgery for Total Hip Arthroplasty (THA)
- SP-CL femur component and Delta TT acetabular component (Active Comparator)
  Interventions: Device: Surgery for Total Hip Arthroplasty (THA)
- SP-CL femoral component and Delta PF acetabular component (Active Comparator)
  Interventions: Device: Surgery for Total Hip Arthroplasty (THA)
- Exeter femoral component and Delta PF acetabular component (Active Comparator)
  Interventions: Device: Surgery for Total Hip Arthroplasty (THA)

INTERVENTIONS:
Device: Surgery for Total Hip Arthroplasty (THA) — THA surgery where four prosthetic components will randomly be inserted. Randomly an Exeter or SP-CL femur component will be combined with randomly a Delta TT or Delta PF acetabular component.

SUMMARY:
What is the intensity of F-PET uptake adjacent to four analyzed hip endoprosthetic components and in healthy femur and acetabulum, 1, 4 and 9 months after surgery?

DETAILED DESCRIPTION:
A clinical study of 32 patients, age 50-69 years, healthy unless osteoarthritis in one hip, randomized in two groups (16 each) plus a reference group of same 32 patient´s contralateral healthy hip.

Intervention will be surgery with a total hip arthroplasty. The four studied endoprosthetic components are:

* Cemented Exeter stem (Stryker Warsaw, USA) with a ceramic 32 mm head and Palacose cement with gentamycin, applied with 3:rd generation cementation technique.
* Uncemented Lubinus SP-CL stem (Waldemar Link, Hamburg, Germany) with a ceramic 32 mm head.
* Uncemented Delta PF cup (Limacorporate spa, Udine, Italy).
* Uncemented fibrous metal Delta TT cup (Limacorporate spa, Udine, Italy). Both cups will have cross linked Ultra-high-molecular-weight polyethylene (UHWMP).

Clinical score, radiography and uptake of Fluoride tracer will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

- patients diagnosed to have unilateral hip osteo arthritis verified by radiography (Charnley group A) aimed for THA at Gävle hospital and accepting to participate in the study.

Exclusion Criteria:

* any systemic disease (other than osteo arthritis) or medication affecting skeleton methabolism

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
FEMUR: to analyze difference in SUV of the 4 upper ROI's (No 1, 7, 8 and 13) analyzed together between the two study groups AND: to analyze SUV of the 4 upper ROI's analyzed together between each femur study group and the reference group | 1 months after surgery
  There are two study groups for femur: cemented and uncemented femur prosthetic components. There is also a femur reference group.
ACETABULUM: to analyze difference in SUV of all 9 ROI's analyzed together between the two study groups (PF and TT), and to analyze SUV of all 9 ROI's analyzed together between each acetabulum prosthetic component study group and the reference group | 1 months after surgery
  There are two study groups for acetabulum: two models of uncemented acetabular prosthetic components. There is also an acetabular reference group.

SECONDARY OUTCOMES:
FEMUR:to analyze difference in SUV for each individual ROI inbetween the cemented and uncemented femur group | 1, 4 and 9 months aftyer surgery
FEMUR: to analyze difference in SUV for each individual ROI between the cemented study group and the reference group. To analyze difference in SUV for each individual ROI between the uncemented study group and the reference group. | 1, 4 and 9 months aftyer surgery
FEMUR:to analyze difference in SUV for each individual ROI between the 3 time points for the cemented group. To analyze difference in SUV for each individual ROI between the 3 time points for the uncemented group. | 1, 4 and 9 months aftyer surgery
FEMUR:to analyze difference in SUV for the 4 upper ROI's (No 1, 7, 8 and 13) analyzed together between the 2 study groups | 4 and 9 months aftyer surgery
FEMUR:to analyze difference in SUV for the 4 upper ROI's analyzed together between each study group and the reference group | 4 and 9 months aftyer surgery
ACETABULUM: to analyze difference in SUV for each individual ROI between the 2 study groups | 1, 4 and 9 months aftyer surgery
ACETABULUM: to analyze difference in SUV for each individual ROI between the two study groups. To analyze difference in SUV for each individual ROI between each of the two study groups and the reference group. | 1, 4 and 9 months aftyer surgery
ACETABULUM: to analyze difference in SUV for each individual ROI for the Delta PF study group between the 3 time points. To analyze difference in SUV for each individual ROI for the Delta TT study group between the 3 time points. | 1, 4 and 9 months aftyer surgery
ACETABULUM: to analyze difference in SUV of all 9 ROI's analyzed together between the two acetabular study groups | 4 and 9 months aftyer surgery
ACETABULUM: to analyze SUV of all 9 ROI's analyzed together between each acetabulum study group and the reference group | 4 and 9 months

OTHER OUTCOMES:
To analyze radiographic difference for each of the four study groups between direct postoperativ and 9 months postoperative radiographs. | Direct postoperative (1-3 days) and 9 months
To analyze clinical score for the four study groups | preoperatively and 9 months postoperatively.
  Merle d Merle d´Aubignè and Postel score

CONTACTS AND LOCATIONS:
Overall Officials: Gösta Ullmark, MD, Principal Investigator — Orthopaedic department Gävle hospital, Gävle, Sweden and Centre for Research & Development Uppsala University/County Council of Gävleborg.
Locations (1):
- Orthopaedic department Gävle hospital, Gävle, Sweden

REFERENCES:
- [Derived] Sotiriou D, Sorensen J, Ullmark G. [18F]-fluoride PET/CT analyses of postoperative bone mineralisation adjacent to femoral stems at THA: a randomised clinical trial. Hip Int. 2025 Nov;35(6):534-542. doi: 10.1177/11207000251372025. Epub 2025 Sep 30. PMID 41025388